CLINICAL TRIAL: NCT05941429
Title: Comparison of Cariostatic Effect of Nano-Silver Fluoride Versus Silver Diamine Fluoride in a Group of Preschool Children
Brief Title: Comparison of Cariostatic Effect of Nano-Silver Fluoride Versus Silver Diamine Fluoride
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lara Abdelmoniem Mohamed, Pediatric dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422021493714
Record Dates: First submitted 2023-06-21; First posted 2023-07-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded study. Participants were blinded towards agents used in the study by using two identical squeezable plastic droppers with tag codes A and B. Also the bio-statistician will be blinded from the meaning of codes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silver Diamine Fluoride (Active Comparator): 38% Silver Diamine Fluoride varnish
  1. the affected tooth will be cleaned by a disposable micro-brush for 30 seconds and then will be dried using cotton gauze sponges.
  2. No excavation will be done to the infected dentin tissue prior to the application of the agent.
  3. Gum will be protected with petroleum jelly, and isolation will be achieved by using cotton rolls.
  4. After isolation, a single drop SDF will be applied into the cavity by using a disposable micro-brush for at least two minutes. Then site of application will be covered with petroleum jelly.
  5. Finally, parents will be instructed that children participating in the trial are not allowed to eat or drink for one hour after application of the agent
  Interventions: Drug: Silver diamine fluoride
- Nano-Silver Fluoride (Experimental): Nano-Silver fluoride varnish preparation
  1. the affected tooth will be cleaned by a disposable micro-brush for 30 seconds and then will be dried using cotton gauze sponges.
  2. No excavation will be done to the infected dentin tissue prior to the application of the agent.
  3. Gum will be protected with petroleum jelly, and isolation will be achieved by using cotton rolls.
  4. After isolation, a single drop NSF will be applied into the cavity by using a disposable micro-brush for at least two minutes. Then site of application will be covered with petroleum jelly.
  5. Finally, parents will be instructed that children participating in the trial are not allowed to eat or drink for one hour after application of the agent
  Interventions: Drug: Nano-Silver Fluoride

INTERVENTIONS:
Drug: Nano-Silver Fluoride — NSF is a varnish which has been introduced as experimental formulation . the laboratory synthesis of NSF was carried out in a nano techonolgy center .
  Other Names: NSF
  Arms: Nano-Silver Fluoride
Drug: Silver diamine fluoride — 38% silver diamine fluoride
  Other Names: SDF
  Arms: Silver Diamine Fluoride

SUMMARY:
This study will be conducted to test the cariostatic effect of Nano Silver Fluoride in a comparison to Silver Diamine Fluoride in a group of preschool children.

DETAILED DESCRIPTION:
Silver Diamine Fluoride has offered a non-invasive and easily performed method to manage dental caries in very young children.Studies shows that SDF has been proven to arrest caries in cavitated lesions and to prevent caries in sound teeth as Fluoride is effective in enhancing the remineralization of dental hard tissue and silver ion acts as an antibacterial agent. However, It was found that silver causes staining to the dental tissues with a black discoloration, which can be considered to be a main drawback specifically, when it is used on anterior teeth. Nano-silver fluoride varnish preparation showed high efficacy in arresting caries progression in primary teeth without causing black discoloration to the tissues.Silver diamine fluoride (SDF) .

Benefits for patient:

1. Non-invasive treatment leading to reduce patient anxiety and stress.
2. No drilling and filling.
3. Protects against further caries progression.

Benefits for the practitioner:

1. Provide alternative treatment options.
2. Pain-free procedure that facilitates child management and saves time.

Benefits for the community:

1. Increasing overall oral health
2. Provides more information by testing new material
3. To provide better service quality.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 3 to 5 years
* clinical diagnosis of active dentinal caries in primary teeth
* Co-operative participants and free of any systemic diseases

Exclusion Criteria:

* Children whose parents refuse to sign consent
* Primary teeth with pulp involvement, pain, mobility, abscess, sinus, fistula; or discoloration related to tooth non-vitality.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
caries lesion activity and severity assessment using Nyvad criteria | baseline
  visual and tactile assessment for caries lesion to evaluate the caries progression using Nyvad classification - score from 0 ( normal enamel translucency and texture ) to 9 (carie lesion with filling )
caries lesion activity and severity assessment using Nyvad criteria | 3 weeks
  visual and tactile assessment for caries lesion to evaluate the caries progression using Nyvad classification - score from 0 ( normal enamel translucency and texture ) to 9 (carie lesion with filling )
caries lesion activity and severity assessment using Nyvad criteria | 6 months
  visual and tactile assessment for caries lesion to evaluate the caries progression using Nyvad classification - score from 0 ( normal enamel translucency and texture ) to 9 (carie lesion with filling )

SECONDARY OUTCOMES:
ICDAS II | baseline
  Detection and assessment of dental caries using ICDAS II - assessment done by photographs - score from 0 ( sound ) to 6 ( Extensive cavity with visible dentin )
ICDAS II | 3 weeks
  Detection and assessment of dental caries using ICDAS II - assessment done by photographs - score from 0 ( sound ) to 6 ( Extensive cavity with visible dentin )
ICDAS II | 6 months
  Detection and assessment of dental caries using ICDAS II - assessment done by photographs - score from 0 ( sound ) to 6 ( Extensive cavity with visible dentin )

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt